CLINICAL TRIAL: NCT04626362
Title: To Determine the Metabolic Polymorphisms of American Cranberries to Prevent UTIs in Susceptible Women Using an Integrated Metabolome-Microbiome Approach
Brief Title: American Cranberries to Prevent UTIs in Susceptible Women
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: IRB202002624
Record Dates: First submitted 2020-10-15; First posted 2020-11-12 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-09

CONDITIONS: Healthy
Keywords: Cranberry; UTI

STUDY DESIGN:
Intervention Model Description: Experimental: Cranberry juice consumption participants will be provided cranberry juice to consume for 21 days Intervention: Other: Cranberry juice Placebo Comparator: Placebo juice consumption participants will be provided placebo juice to consume for 21 days Intervention: Other: Placebo juice
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Cranberry juice consumption (Experimental): Participants will be provided with cranberry juice to consume for 4 days after 10 10-day run-in period.
  Interventions: Other: Cranberry juice

INTERVENTIONS:
Other: Cranberry juice — Cranberry juice cocktail is a product of Ocean Spray Cranberries, Inc.

SUMMARY:
The investigator's pre-preliminary study showed that the urine from a portion of study participants had anti-adhesion activity. The investigators propose that UTI susceptible women can be divided into responders and non-responders depending on whether cranberry intake increases anti-adhesion activity of their urine.

DETAILED DESCRIPTION:
The American cranberries (Vaccinium macrocarpon) have been consumed for centuries to prevent urinary tract infections (UTIs), which affect 50% of women in their lifetime. However, NIH-funded clinical trials of cranberries on UTI in the last 20 years yielded conflicting results, but the reasons are unknown. About 90% of UTIs are initiated by adhesion of uropathogenic E. coli on urinary tract epithelia. It was reported that human urine after cranberry intake inhibited the adhesion of E. coli. A-type procyanidins and xyloglucans are the presumed bioactives in cranberries; however, none of these compounds are absorbable in the small intestine. They are degraded by microbes in the colon. The pre-preliminary study showed that the urine from a portion of study participants had anti-adhesion activity, suggesting there are polymorphisms in humans' ability to metabolize cranberry bioactives. The investigators propose that UTI susceptible women can be divided into responders and non-responders depending on whether cranberry intake increases anti-adhesion activity of their urine.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women participants
* BMI 18.5-29.9 kg/m2
* At least 110 pounds in weight

Exclusion Criteria:

* BMI≥ 30 kg/m2
* Pregnancy and breast-feeding
* Smoking, frequent alcohol use
* History of any clinically important disorder that may interfere with interpretation of the results,
* Intake of medication that might influence the outcome of the study

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — UTI predominantly affect women and is rare in men.
Enrollment: 55 (Actual)
Dates: Start 2021-02-02 (Actual); Primary Completion 2026-08-20 (Estimated); Study Completion 2026-08-20 (Estimated)

PRIMARY OUTCOMES:
baseline urinary anti-adhesion index | day 9 and 10
  During the 10-day run-in period, all the participants will be given a list of foods to avoid, including cranberries, blueberries, grapes, apples, plums, chocolate, and green tea. Two self-collected baseline urine samples will be provided by participants on the mornings of days 9 and 10. Anti-adhesion activity of urine against E coli will be assessed using a fluorescent method.

SECONDARY OUTCOMES:
Urinary anti-adhesion index after four days of cranberry juice intake | after drinking cranberry juice for 4 days
  After urine collection in the last two days of the run-in period, participants will maintain their dietary restriction for an additional 2-7 days and allow the anti-adhesion activity of baseline urine to be tested. Afterward, part of the participants will be selected to consume cranberry juice for four days. Each participant drank two bottles of cranberry cocktail containing 27% juice per day. A post-consumption urine sample will be self-collected by each participant on the morning of day 5. Anti-adhesion activity of urine against E coli will be assessed using a fluorescent method.

CONTACTS AND LOCATIONS:
Overall Officials: Liwei Gu, PhD, Principal Investigator — University of Florida; Yavuz Yagiz, PhD, Study Director — University of Florida
Locations (1):
- Food Science and human nutrition department at University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No